CLINICAL TRIAL: NCT06116292
Title: Impact of the Implementation of a Telemedicine Program on Patients Diagnosed with Asthma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, Héctor Cabrerizo Carreño, Principal Investigator, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TAPR-578/24
Record Dates: First submitted 2023-10-22; First posted 2023-11-03 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Asthma; Telemedicine; Adherence, Treatment; Quality of Life; Control
Keywords: Asthma; Telemedicine; Asthma Control; Quality of Live; Adherence, Treatment
MeSH Terms: conditions — Asthma; Treatment Adherence and Compliance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mobile application ESTOI for Asthmatic patients (Experimental): The intervention group will receive the usual care, in addition to having access to the ESTOI application.
  Interventions: Device: The mobile application ESTOI for Asthmatic patients
- Standard of care (No Intervention): The intervention group will receive the usual care

INTERVENTIONS:
Device: The mobile application ESTOI for Asthmatic patients — The mobile application ESTOI have various sections that can be managed and customized by the researchers to meet each patient's needs:
  1. SYMPTOM CONTROL, it will record the ACT, TAI, the number of exacerbations, weight, and, depending on the case, symptom control for comorbidities.
  2. RECOMMENDATIONS, it will provide patients with information needed to understand their condition, how to control it, and what to do in case of worsening symptoms.
  3. YOUR TREATMENT, it will display personalized and update information about the patient's current asthma medication, including dosages and frequencies. There will be explanatory videos on how to administer the therapy and includes an action plan.
  4. PEAK FLOW, the patient can record measurements using a Peak Flow Meter at home.
  5. NUTRITIONAL PLAN, it will provide a daily dietary guide to enable individuals to adapt these tools and recommendations to their specific needs.
  6. MESSAGING, it is a bidirectional contact area.
  Arms: Mobile application ESTOI for Asthmatic patients

SUMMARY:
Introduction: Asthma is one of the most common chronic respiratory diseases worldwide. Despite the extensive knowledge of the condition and available therapeutic options, severe asthmatic patients have poor disease control in 50% of cases.

Objective: To assess the impact of implementing a mobile application (ESTOI) in patients diagnosed with asthma on disease control, treatment adherence, and perceived quality of life.

Methodology: A 52-week randomized clinical trial involving asthma patients receiving care at a highly specialized hospital in Spain. A total of 108 patients will be included and divided into two groups. The intervention group will receive more comprehensive monitoring than usual, including access to the ESTOI application. The Asthma Control Test (ACT) questionnaire will be used as the primary assessment variable. Other variables to be studied include the Inhaler Adherence Test (TAI), the number of exacerbations, peak expiratory flow, exhaled nitric oxide examination, hospital anxiety and depression scale, asthma quality of life questionnaire, forced spirometry parameters (FVC, FEV1, and reversibility), and analytical parameters (eosinophilia and IgE).

DETAILED DESCRIPTION:
Design: A 52-week randomized clinical trial will be conducted, using a single-blind approach, in patients with asthma. There will be two study arms: the control cohort will receive standard care, while the intervention group will also have access to the mobile application (ESTOI).

Setting and Subjects: The study will take place in the pulmonology department of Bellvitge University Hospital in Barcelona, during the years 2024-2026.

Procedure and Instruments: The project will be structured into three visits. During the first visit, all participants will be seen by the pulmonologist at our center for asthma classification, inhaler updates, and requests for additional tests. Subsequently, the control group will receive health education (provided by the asthma specialist nurse) regarding their condition, treatment plan, signs of alarm, action plan, and a review of asthma triggers. On the other hand, intervention group patients, in addition to health education, will be introduced to the ESTOI application database and provided access to the patient portal, where patients will find all the necessary information on asthma management. Both groups will receive a Peakflow meter and instructions on its use and record-keeping.

A nurse will be responsible for managing and monitoring the patients using the application. Patients will also schedule and review the medical records of all patients included in the study and review the data collection notebooks and informed consents. The asthma specialist nurse will be responsible for conducting the questionnaires, collecting data for the Case Report Form (CRF), performing laboratory tests, and conducting respiratory functional tests.

During the three study visits, all included patients will complete the study questionnaires: Asthma Control Test (ACT), Inhaler Adherence Test (TAI), Asthma Quality of Life Questionnaire (AQLQ), and the Hospital Anxiety and Depression Scale (HAD). Afterward, the electronic history of medication dispenses will be reviewed, exhaled nitric oxide (FeNO) will be measured, a spirometry test with bronchodilator response, a control blood test, and an on-site measurement of Peak Expiratory Flow (PEF) using the Peakflow meter will be conducted.

At the end of the first visit, all participants will be scheduled for the next visit and provided with a contact phone number in case the patients have any questions or issues.

Upon completion of the third visit, the intervention group will be given a satisfaction questionnaire for having used the application."

All relevant study data will be recorded in each patient's data collection notebook for subsequent analysis. These notebooks will be stored at the center in a locked room accessible only to the research team. Sociodemographic variables will be collected by the asthma unit nurse during the first study visit.

Information about the current state of asthma will be obtained through questionnaires, respiratory functional tests, laboratory tests, and a review of the patient's medical history.

Data Analysis: Continuous variables will be expressed as mean and standard deviation in case of a normal distribution, and as median and interquartile range in case of a non-normal distribution. Qualitative variables will be presented as frequencies and percentages. For the comparison of continuous variables, analysis of variance (ANOVA) or the Kruskal-Wallis test will be used. The chi-square test will be performed for the analysis of the primary outcome variable. Stepwise logistic regression models will be used to select the subgroup of parameters significantly associated with poor asthma control. A priori, the factors included in the analysis will be age, asthma duration, education level, BMI, smoking, environmental exposure, pre-BD FEV1, post-BD FEV1, FeNO, blood eosinophilia, general and specific blood IgE levels, ACT, TAI, HAD, AQLQ, the number of exacerbations, and control of comorbidities affecting asthma (GERD, rhinitis, polyps, overweight/obesity, and smoking). Statistical significance will be assumed at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years with a diagnosis of asthma based on GEMA 5.2 2022.
* Patients seen in the pulmonology service of the center.
* Patients who have not previously received asthma education.
* Capable of giving signed informed consent.

Exclusion Criteria:

* Patient who does not have a mobile device with Android or IOS system.
* Lack of minimum technological knowledge for the use of the application (ESTOI).
* People who are participating or have participated in a clinical trial in the last 6 months.
* Patients diagnosed with other respiratory diseases except for obstructive sleep apnea (OSA), Asthma-COPD overlap syndrome (ACOS).
* Patients with palliative or severe chronic illnesses that limit their life expectancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Asthma Control Test (ACT) | Visit 1 (week 0), visit 2 (week 26) and visit 3 (week 52)
  ACT is a 5-item questionnaire that assesses the level of control of asthma symptoms during the previous 4 weeks. The results range from 5 to 25, where higher results indicate better control of the disease and low results indicate worse control. Results between 20 and 25 are established as good control, partial control between 16 and 19, and poor control less than 15.
Number of exacerbations | Visit 1 (week 0), visit 2 (week 26) and visit 3 (week 52).
  In asthma an exacerbation is considered a worsening of asthma symptoms that requires medical intervention and has at least 1 of the following 3 elements listed below for at least 2 consecutive days: Worsening of asthma signs/symptoms (dyspnea, wheezing, nocturnal awakenings, or chest tightness), increased use of rescue medication or deterioration of lung function.
Peak Expiratory Flow (PEF) | Visit 1 (week 0), visit 2 (week 26) and visit 3 (week 52)
  It will be use the PEF to to know the current lung status and the degree of asthma control. At each visit, a PEF measurement will be performed. A good control will be considered when the results obtained in PEF are greater than 80% compared to the patient's personal best.
Forced expiratory volume in one second (FEV1) | Visit 1 (week 0), visit 2 (week 26) and visit 3 (week 52)
  It will be use the FEV1 to to know the current lung status and the degree of asthma control. At each visit, a spirometry will be performed. A good control will be considered when the results obtained in these tests are greater than 80% compared to the patient's personal best or the theoretical value or zscore (-1.64).

SECONDARY OUTCOMES:
Test of the Adherence to Inhalers (TAI). | Visit 1 (week 0), visit 2 (week 26) and visit 3 (week 52)
  TAI is a 12-item questionnaire that assesses adherence to inhalers for patients with Asthma or COPD. Thus, if the healthcare professional only wants to assess adherence and its intensity, patients should use the 10-item TAI. If he also wants to assess the type of non-compliance, he can use the 12-item TAI. The type or pattern of non-compliance will be assessed as follows: Items 1 to 5 assess "erratic" non-compliance (score between 5 and 25), items 6 to 10 assess "deliberate" non-compliance (score between 5 and 25) and items 11 and 12 assess "unconscious" non-compliance (score between 2 and 4).
Electronic history of medication dispenses | Visit 1 (week 0), visit 2 (week 26) and visit 3 (week 52)
  In order to assess treatment adherence, the electronic history of medication dispenses will be reviewed. The investigator could see how many times the patient draws his treatment each month. This will help to observe if treatment compliance is optimal, but it should be used in conjunction with the TAI to ensure the results.
Asthma Quality of Life Questionnaire (AQLQ) | Visit 1 (week 0), visit 2 (week 26) and visit 3 (week 52)
  AQLQ is a 32-item questionnaire that assesses the quality of life of patients with asthma. Covers 4 dimensions (breathlessness, mood, social limitation and worrying). Answers are given on a scale of 7 points, where 1 = maximum limitation and 7 = absence of limitation. The questionnaire provides an overall score, which is the average for all items, and a score for each dimension, which is the average of the corresponding items.
The Hospital Anxiety and Depression Scale (HADS) | Visit 1 (week 0), visit 2 (week 26) and visit 3 (week 52)
  HADS is a questionnaire for detecting affective disorders in hospital settings with outpatients. Is frequently used to evaluate populations with chronic diseases. It consists of 14 items. Odd items configure the subscale of anxiety and its response scale is scored from 3 to 0. The pairs make up the depression subscale and are scored from 0 to 3. The total score on each subscale is obtained by adding those of the corresponding items, with each range from 0 to 21. In both cases, the higher the score, the higher the level of anxiety or depression.

CONTACTS AND LOCATIONS:
Overall Officials: Héctor Cabrerizo Carreño, M.N, Principal Investigator — Hospital Universitari de Bellvitge; Mariana M Muñoz, M.D., Study Director — Hospital Universitari de Bellvitge
Locations (1):
- Bellvitge University Hospital, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
At the moment, the investigator team have not yet decided whether to make all the patient data collected in this study available to other researchers. If the investigator do choose to share the data, it would include sociodemographic information, data collected from the questionnaires administered throughout the study, results obtained from pulmonary function tests (also obtained through the mobile app), the number of app logins, video views, questionnaire response rates, peak expiratory flow (PEF) records, the number of consultations with healthcare professionals through the app, and analytical parameters. When the results have been published, the principal investigator will consider whether it would be beneficial to present all of these findings.

REFERENCES:
- [Background] GBD 2015 Chronic Respiratory Disease Collaborators. Global, regional, and national deaths, prevalence, disability-adjusted life years, and years lived with disability for chronic obstructive pulmonary disease and asthma, 1990-2015: a systematic analysis for the Global Burden of Disease Study 2015. Lancet Respir Med. 2017 Sep;5(9):691-706. doi: 10.1016/S2213-2600(17)30293-X. Epub 2017 Aug 16. PMID 28822787
- [Background] Plaza V, Quirce S, Delgado J, Martinez Moragon E, Perez de Llano L; Grupo multidisciplinar de expertos "Asmaforum". [Multidisciplinary expert discussion. Uncontrolled asthma: causes, consequences and possible solutions]. An Sist Sanit Navar. 2016 Nov 21;39(3):357-370. doi: 10.23938/ASSN.0233. Spanish. PMID 28032871
- [Background] Rabe KF, Adachi M, Lai CK, Soriano JB, Vermeire PA, Weiss KB, Weiss ST. Worldwide severity and control of asthma in children and adults: the global asthma insights and reality surveys. J Allergy Clin Immunol. 2004 Jul;114(1):40-7. doi: 10.1016/j.jaci.2004.04.042. PMID 15241342
- [Background] Quirce S, Plaza V, Picado C, Vennera M, Casafont J. Prevalence of uncontrolled severe persistent asthma in pneumology and allergy hospital units in Spain. J Investig Allergol Clin Immunol. 2011;21(6):466-71. PMID 21995180
- [Background] Almonacid Sanchez C, Blanco Aparicio M, Dominguez Ortega J, Giner Donaire J, Molina Paris J, Sanchez Marcos N, Plaza V. [Multidisciplinary Consensus for the Monitoring and Control of Asthma Through Telemedicine. The COMETA Project]. Open Respir Arch. 2021 Apr 19;3(2):100098. doi: 10.1016/j.opresp.2021.100098. eCollection 2021 Apr-Jun. Spanish. PMID 37497073
- [Background] Marcano Belisario JS, Huckvale K, Greenfield G, Car J, Gunn LH. Smartphone and tablet self management apps for asthma. Cochrane Database Syst Rev. 2013 Nov 27;2013(11):CD010013. doi: 10.1002/14651858.CD010013.pub2. PMID 24282112
- [Background] Hollenbach JP, Cushing A, Melvin E, McGowan B, Cloutier MM, Manice M. Understanding clinicians' attitudes toward a mobile health strategy to childhood asthma management: A qualitative study. J Asthma. 2017 Sep;54(7):754-760. doi: 10.1080/02770903.2016.1263649. Epub 2016 Nov 23. PMID 27880049
- [Background] Munteanu LA, Frandes M, Timar B, Tudorache E, Fildan AP, Oancea C, Tofolean DE. The efficacy of a mobile phone application to improve adherence to treatment and self-management in people with chronic respiratory disease in Romanian population - a pilot study. BMC Health Serv Res. 2020 May 27;20(1):475. doi: 10.1186/s12913-020-05340-0. PMID 32460752
- [Background] Guan Z, Sun L, Xiao Q, Wang Y. Constructing an assessment framework for the quality of asthma smartphone applications. BMC Med Inform Decis Mak. 2019 Oct 15;19(1):192. doi: 10.1186/s12911-019-0923-8. PMID 31615493
- [Background] Farzandipour M, Nabovati E, Heidarzadeh Arani M, Akbari H, Sharif R, Anvari S. Enhancing Asthma Patients' Self-Management through Smartphone-Based Application: Design, Usability Evaluation, and Educational Intervention. Appl Clin Inform. 2019 Oct;10(5):870-878. doi: 10.1055/s-0039-1700866. Epub 2019 Nov 13. PMID 31724144
- [Background] Morrison D, Wyke S, Agur K, Cameron EJ, Docking RI, Mackenzie AM, McConnachie A, Raghuvir V, Thomson NC, Mair FS. Digital asthma self-management interventions: a systematic review. J Med Internet Res. 2014 Feb 18;16(2):e51. doi: 10.2196/jmir.2814. PMID 24550161
- [Background] Thomas M, Kay S, Pike J, Williams A, Rosenzweig JR, Hillyer EV, Price D. The Asthma Control Test (ACT) as a predictor of GINA guideline-defined asthma control: analysis of a multinational cross-sectional survey. Prim Care Respir J. 2009 Mar;18(1):41-9. doi: 10.4104/pcrj.2009.00010. PMID 19240948
- [Background] Plaza V, Fernandez-Rodriguez C, Melero C, Cosio BG, Entrenas LM, de Llano LP, Gutierrez-Pereyra F, Tarragona E, Palomino R, Lopez-Vina A; TAI Study Group. Validation of the 'Test of the Adherence to Inhalers' (TAI) for Asthma and COPD Patients. J Aerosol Med Pulm Drug Deliv. 2016 Apr;29(2):142-52. doi: 10.1089/jamp.2015.1212. Epub 2015 Jul 31. PMID 26230150
- [Background] Perpina M, Belloch A, Pascual LM, de Diego A, Compte L. [The quality of life in asthma: an evaluation of the AQLQ questionnaire for its use on a Spanish population. Asthma Quality of Life Questionnaire]. Arch Bronconeumol. 1995 May;31(5):211-8. doi: 10.1016/s0300-2896(15)30926-1. Spanish. PMID 7788082
- [Background] Reddel HK, Marks GB, Jenkins CR. When can personal best peak flow be determined for asthma action plans? Thorax. 2004 Nov;59(11):922-4. doi: 10.1136/thx.2004.023077. PMID 15516464
- [Background] Pellegrino R, Viegi G, Brusasco V, Crapo RO, Burgos F, Casaburi R, Coates A, van der Grinten CP, Gustafsson P, Hankinson J, Jensen R, Johnson DC, MacIntyre N, McKay R, Miller MR, Navajas D, Pedersen OF, Wanger J. Interpretative strategies for lung function tests. Eur Respir J. 2005 Nov;26(5):948-68. doi: 10.1183/09031936.05.00035205. No abstract available. PMID 16264058
- [Background] Lu Z, Huang W, Wang L, Xu N, Ding Q, Cao C. Exhaled nitric oxide in patients with chronic obstructive pulmonary disease: a systematic review and meta-analysis. Int J Chron Obstruct Pulmon Dis. 2018 Aug 30;13:2695-2705. doi: 10.2147/COPD.S165780. eCollection 2018. PMID 30214187
- [Background] Schatz M, Kosinski M, Yarlas AS, Hanlon J, Watson ME, Jhingran P. The minimally important difference of the Asthma Control Test. J Allergy Clin Immunol. 2009 Oct;124(4):719-23.e1. doi: 10.1016/j.jaci.2009.06.053. Epub 2009 Sep 19. PMID 19767070
- [Background] Kolmodin MacDonell K, Naar S, Gibson-Scipio W, Lam P, Secord E. The Detroit Young Adult Asthma Project: Pilot of a Technology-Based Medication Adherence Intervention for African-American Emerging Adults. J Adolesc Health. 2016 Oct;59(4):465-71. doi: 10.1016/j.jadohealth.2016.05.016. Epub 2016 Jul 27. PMID 27475032
- [Background] Patel MR, Song PX, Sanders G, Nelson B, Kaltsas E, Thomas LJ, Janevic MR, Hafeez K, Wang W, Wilkin M, Johnson TR, Brown RW. A randomized clinical trial of a culturally responsive intervention for African American women with asthma. Ann Allergy Asthma Immunol. 2017 Feb;118(2):212-219. doi: 10.1016/j.anai.2016.11.016. Epub 2016 Dec 27. PMID 28034579
- [Background] Kim MY, Lee SY, Jo EJ, Lee SE, Kang MG, Song WJ, Kim SH, Cho SH, Min KU, Ahn KH, Chang YS. Feasibility of a smartphone application based action plan and monitoring in asthma. Asia Pac Allergy. 2016 Jul;6(3):174-80. doi: 10.5415/apallergy.2016.6.3.174. Epub 2016 Jul 28. PMID 27489790
- [Background] Zairina E, Abramson MJ, McDonald CF, Li J, Dharmasiri T, Stewart K, Walker SP, Paul E, George J. Telehealth to improve asthma control in pregnancy: A randomized controlled trial. Respirology. 2016 Jul;21(5):867-74. doi: 10.1111/resp.12773. Epub 2016 Mar 31. PMID 27037722
- [Background] Pool AC, Kraschnewski JL, Poger JM, Smyth J, Stuckey HL, Craig TJ, Lehman EB, Yang C, Sciamanna CN. Impact of online patient reminders to improve asthma care: A randomized controlled trial. PLoS One. 2017 Feb 3;12(2):e0170447. doi: 10.1371/journal.pone.0170447. eCollection 2017. PMID 28158200
- [Background] Khusial RJ, Honkoop PJ, Usmani O, Soares M, Simpson A, Biddiscombe M, Meah S, Bonini M, Lalas A, Polychronidou E, Koopmans JG, Moustakas K, Snoeck-Stroband JB, Ortmann S, Votis K, Tzovaras D, Chung KF, Fowler S, Sont JK; myAirCoach study group. Effectiveness of myAirCoach: A mHealth Self-Management System in Asthma. J Allergy Clin Immunol Pract. 2020 Jun;8(6):1972-1979.e8. doi: 10.1016/j.jaip.2020.02.018. Epub 2020 Mar 3. PMID 32142961
- [Background] Cao Y, Lin SH, Zhu D, Xu F, Chen ZH, Shen HH, Li W. WeChat Public Account Use Improves Clinical Control of Cough-Variant Asthma: A Randomized Controlled Trial. Med Sci Monit. 2018 Mar 14;24:1524-1532. doi: 10.12659/msm.907284. PMID 29536984
- [Background] Prabhakaran L, Chun Wei Y. Effectiveness of the eCARE programme: a short message service for asthma monitoring. BMJ Health Care Inform. 2019 Jun;26(1):e100007. doi: 10.1136/bmjhci-2019-100007. PMID 31201202
- [Background] Nemanic T, Sarc I, Skrgat S, Flezar M, Cukjati I, Marc Malovrh M. Telemonitoring in asthma control: a randomized controlled trial. J Asthma. 2019 Jul;56(7):782-790. doi: 10.1080/02770903.2018.1493599. Epub 2018 Sep 5. PMID 30063840
- [Background] Ahmed S, Ernst P, Bartlett SJ, Valois MF, Zaihra T, Pare G, Grad R, Eilayyan O, Perreault R, Tamblyn R. The Effectiveness of Web-Based Asthma Self-Management System, My Asthma Portal (MAP): A Pilot Randomized Controlled Trial. J Med Internet Res. 2016 Dec 1;18(12):e313. doi: 10.2196/jmir.5866. PMID 27908846
- [Background] Koufopoulos JT, Conner MT, Gardner PH, Kellar I. A Web-Based and Mobile Health Social Support Intervention to Promote Adherence to Inhaled Asthma Medications: Randomized Controlled Trial. J Med Internet Res. 2016 Jun 13;18(6):e122. doi: 10.2196/jmir.4963. PMID 27298211
- [Background] Chongmelaxme B, Lee S, Dhippayom T, Saokaew S, Chaiyakunapruk N, Dilokthornsakul P. The Effects of Telemedicine on Asthma Control and Patients' Quality of Life in Adults: A Systematic Review and Meta-analysis. J Allergy Clin Immunol Pract. 2019 Jan;7(1):199-216.e11. doi: 10.1016/j.jaip.2018.07.015. Epub 2018 Jul 25. PMID 30055283
- [Derived] Cabrerizo-Carreno H, Munoz-Esquerre M, Santos Perez S, Romero-Ortiz AM, Fabrellas N, Guix-Comellas EM. Impact of the implementation of a telemedicine program on patients diagnosed with asthma. BMC Pulm Med. 2024 Jan 13;24(1):32. doi: 10.1186/s12890-024-02843-y. PMID 38216971
- See also: Global burden of 369 diseases and injuries in 204 countries and territories, 1990-2019: a systematic analysis for the Global Burden of Disease Study 2019 — https://linkinghub.elsevier.com/retrieve/pii/S0140673620309259
- See also: Gina Main report 2022 — https://ginasthma.org/gina-reports/
- See also: Difficult to control asthma: predisposing and aggravating factors — http://www.elsevier.es/es-revista-revista-patologia-respiratoria-318-articulo-asma-control-dificil-factores-predisponentes-X1576989511020186
- See also: Anxiety scale HADS — https://www.redalyc.org/journal/1339/133959841009/133959841009.pdf
- See also: Random. org — http://www.random.org/strings/